CLINICAL TRIAL: NCT00300300
Title: Anterior Cruciate Ligament Reconstruction: Comparison of Patellar With Hamstring Tendon Using a Computer-assisted Versus a Conventional Surgical Technique.
Brief Title: Anterior Cruciate Ligament (ACL) Reconstruction Using Different Grafts and Surgical Techniques
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study temporarily suspended until funding can be secured.
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. David Bardana, Principal Investigator, Queen's University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Bard0105
Record Dates: First submitted 2006-03-06; First posted 2006-03-08 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: ACL computer-assisted surgery graft
MeSH Terms: interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (No Intervention): applying a patellar graft using conventional surgical technique.
- 2 (No Intervention): applying a hamstring graft using conventional surgical technique.
- 3 (Experimental): applying a patellar graft using a computer-assisted surgy technique.
  Interventions: Procedure: Computer-assisted surgery
- 4 (Experimental): hamstring graft CAOS
  Interventions: Procedure: Computer-assisted surgery

INTERVENTIONS:
Procedure: Computer-assisted surgery — no description
  Arms: 3; 4

SUMMARY:
ACL reconstruction in the Division of Orthopaedic surgery at Queen's is currently being performed arthroscopically assisted. The resultant function of the reconstructed ligament is greatly influenced by the placement of the transosseous tunnels, which are tunnels in the bones through which the grafts pass. Presently the placement of the tunnels is being judged from arthroscopically identified anatomical landmarks within the joint. The result is incidence rates of misplaced tunnels as high as 40%. Computer assisted tunnel placement would aid in the correction and reproducibility of anatomic tunnel placement. The objective of this study is to conduct a prospective, randomized trial comparing clinical and radiographic outcomes in subjects who receive either a patella or hamstring tendon graft to reconstruct a chronic tear of the anterior cruciate ligament. All subjects will be further randomized into a computer-assisted or a conventional arthroscopic surgical group to allow investigators to compare the precision and accuracy of tunnel placement between these surgical approaches. The main question under investigation is: does the increased accuracy of computer-assisted surgery make a clinical difference to the laxity of the reconstructed knee, and is the laxity further influenced by the type of tendon graft received?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a chronic unilateral rupture of the anterior cruciate ligament
* Aged 18-40

Exclusion Criteria:

* Acute injury of the ACL (interval between the injury and operation is < 30 days).
* Other ligament tears and/or operation on the operative knee (with the exception of a previous meniscectomy).
* Injury of the contralateral knee.
* Degenerative changes of the articular cartilage (grade III or IV changes according to the Outerbrige classification system)
* Complaints of patellofemoral symptoms
* Patient is pregnant
* Inability to complete 2-year follow-up

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2009-09; Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
The main outcome under investigation is knee laxity as reflected by graft tension. | 2 years

SECONDARY OUTCOMES:
Other outcomes of interest include graft isometry, position and size as well as knee pain, stiffness, function, and range of motion. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Davide Bardana, MD, Principal Investigator — Queen's University (faculty)
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada